CLINICAL TRIAL: NCT03993873
Title: A Phase 1/2 of Study of the Safety, Tolerability, Pharmacokinetics, and Efficacy of TPX-0022 in Adult Subjects With Locally Advanced or Metastatic NSCLC, Gastric Cancer, or Solid Tumors Harboring Genetic Alterations in MET
Brief Title: Study of TPX-0022 in Patients With Advanced NSCLC, Gastric Cancer or Solid Tumors Harboring Genetic Alterations in MET
Acronym: SHIELD-1
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Turning Point Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA177-1036; CA177-1036 (Other: Bristol-Myers Squibb Protocol ID); TPX-0022-01 (Other: Turning Point Therapeutics Protocol ID)
Record Dates: First submitted 2019-06-13; First posted 2019-06-21 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Advanced Solid Tumor; Metastatic Solid Tumors; MET Gene Alterations
Keywords: Non Small Cell Lung; Non Small Cell Lung Cancer; Non-small cell lung cancer; NSCLC; TPX-0022; EGFR wild-type (wt); advanced non-small cell lung cancer; advanced/metastatic disease; Non-small cell lung carcinoma (NSCLC); treatment of lung cancer after first metastasis; treatment of gastric cancer after first metastasis; treatment of hepatocellular cancer after first metastasis; lung cancer; lung adenocarcinoma; Non small cell lung carcinoma; MET exon 14 deletion; MET exon 14 skipping; MET exon 14 mutation; MET mutation; MET amplification; MET inhibitor; MET dysregulation; MET activation; MET signaling; MET pathway; MET fusion; gastric cancer; hepatocellular cancer; SRC; CSF1R; cancer; first in human
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis; Lung Neoplasms; Adenocarcinoma of Lung; Stomach Neoplasms; Liver Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Phase 1 elzovantinib (Experimental): The dose-escalation part of the study will determine the safety, tolerability, MTD, and RP2D of elzovantinib.
  The dose-expansion part of the study will determine the safety, tolerability, PK, and preliminary efficacy in specific cohorts.
  Dose expansion cohorts: Cohort I (NSCLC, METΔex14, treatment Naive) Enrollment Closed; Cohort II (NSCLC with METΔex14, MET therapy pre-treated) Enrollment closed; Cohort III (MET amplified NSCLC, GCN≥10); Cohort IV (MET amplified GI cancer GC/GEJ, CRC/HCC, GCN≥10); Cohort V (NSCLC or GI MET amplified, GCN≥5 and < 10); Cohort VI (Solid tumors with MET fusions, or oncogenic MET mutations or MET amplified other than GI/NSCLC
  Interventions: Drug: elzovantinib (TPX-0022)

INTERVENTIONS:
Drug: elzovantinib (TPX-0022) — Oral elzovantinib (TPX-0022) capsules

SUMMARY:
A phase 1/2, first-in-human, open-label study of the safety, tolerability, PK, and efficacy of the novel MET/CSF1R/SRC inhibitor TPX-0022 in adult subjects with advanced or metastatic NSCLC, Gastric Cancer, or solid tumors harboring genetic alterations in MET. (SHIELD-I)

DETAILED DESCRIPTION:
Dose Escalation: To evaluate the overall safety profile of TPX-0022, single and multiple dose PK profiles and preliminary efficacy in adults subjects with advanced solid tumors harboring genetic alterations in MET.

Dose Expansion: To evaluate the preliminary efficacy and overall safety profile of TPX-0022 at the RP2D in defined cohorts of adult subjects in NSCLC, Gastric Cancer and advanced solid tumors harboring genetic alterations in MET.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 (or age ≥ 20 as required by local regulation).
2. Histological or cytological confirmation of advanced/metastatic MET exon 14 skipping mutation (METΔex14) NSCLC, MET amplified NSCLC, or MET amplified gastric cancers as determined by FISH, qPCR or NGS by local liquid biopsy or tissue, solid tumors with MET fusions or oncogenic MET mutations or MET amplified other than GI/NSCLC.
3. ECOG performance status ≤ 1.
4. Existence of measurable or evaluable disease (according to Response evaluation criteria in solid tumors [RECIST v1.1] criteria).
5. Subjects with asymptomatic primary CNS tumors or brain metastases are eligible for the study if they meet protocol specified criteria.
6. Adequate organ function.
7. Life expectancy ≥ 12 weeks.

Exclusion Criteria:

1. Locally advanced solid tumor that is a candidate for curative treatment through radical surgery and/or radiotherapy, or chemotherapy.
2. Presence or history of any other primary malignancy within the past 3 years other than a history of adequately treated basal or squamous cell carcinoma of the skin, or any adequately treated in situ carcinoma.
3. Major surgery within four weeks of the start of therapy.
4. Additional exclusion criteria for subjects with NSCLC with MET alterations: known oncogene mutations (eg, ALK, ROS1, KRAS, EGFR, etc.) for which there are approved therapies.
5. Additional exclusion criteria for subjects with HCC with MET alterations: liver dysfunction greater than Child-Pugh Class A.
6. Clinically significant cardiovascular disease (either active or within six months before enrollment): myocardial infarction, unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure (New York Heart Association Classification Class ≥ II), cerebrovascular accident or transient ischemic attack, symptomatic bradycardia, requirement for anti-arrhythmic medication. Ongoing cardiac dysrhythmias of CTCAE version 5.0 grade ≥ 2.
7. Any of the following cardiac criteria:

   * Mean resting corrected QT interval (ECG interval measured from the onset of the QRS complex to the end of the T wave) for heart rate (QTc) > 470 msec obtained from three ECGs, using the screening clinic ECG machine-derived QTc value
   * Any clinically important abnormalities in rhythm, conduction, or morphology of resting ECG (e.g., complete left bundle branch block, third degree heart block, second degree heart block, PR interval > 250 msec)
   * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, congenital long QT syndrome, family history of long QT syndrome, or any concomitant medication known to prolong the QT interval
8. Known clinically significant active infections not controlled with systemic treatment (bacterial, fungal, viral including HIV positivity).
9. Peripheral neuropathy ≥ Grade 2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2019-09-05 (Actual); Primary Completion 2024-01-08 (Actual); Study Completion 2027-03-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of first cycle dose-limiting toxicities (DLTs) of elzovantinib | Within 28 days of the first elzovantinib dose for each patient
  Evaluate the safety and tolerability of elzovantinib
Define the Recommended Phase 2 Dose | Approximately 48 months
  Determine the maximum tolerated dose (MTD) and/or Recommended Phase 2 Dose (RP2D) of elzovantinib

SECONDARY OUTCOMES:
Adverse events (AEs) | Approximately 48 months
  Evaluate the overall safety profile of elzovantinib
Cmax (maximum plasma concentration) of elzovantinib | Up to 72 hours post-dose
  Evaluate the maximum plasma concentration of elzovantinib
AUC (area under plasma concentration time curve) of elzovantinib | Up to 72 hours post-dose
  Evaluate the AUC of elzovantinib
Cmax (maximum plasma concentration) of TPX-0022 under different food intake conditions | Up to 72 hours post-dose
  Determine the effect of food (specifically, a high-fat, high-calorie meal) on the single-dose PK (Cmax) of elzovantinib at the RP2D
AUC (area under plasma concentration time curve) of elzovantinib under different food intake conditions | Up to 72 hours post-dose
  Determine the effect of food (specifically, a high-fat, high-calorie meal) on the single-dose PK (AUC) of elzovantinib at the RP2D
Preliminary Objective Response Rate (ORR) | Approximately 48 months
  Determine the preliminary objective response rate (ORR) by Blinded Independent Central Review (BICR) of elzovantinib
Clinical benefit rate (CBR) | Approximately 48 months
  Determine the CBR of elzovantinib
Time to response (TTR) | Approximately 48 months
  Determine the TTR of elzovantinib
Duration of Response (DOR) | Approximately 48 months
  Determine the DOR of elzovantinib
Progression free survival (PFS) | Approximately 48 months
  Determine the PFS of elzovantinib
Intracranial tumor response | Approximately 48 months
  Determine the intracranial tumor response in subjects with measurable brain metastases, as determined by BICR
Overall survival (OS) | Approximately 48 months
  Determine efficacy and safety of elzovantinib

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (24):
- United States (12):
  - Local Institution - 2102, La Jolla, California
  - Local Institution - 2108, Orange, California
  - Local Institution - 2105, Denver, Colorado
  - Local Institution - 2111, Chicago, Illinois
  - Local Institution - 2107, Boston, Massachusetts
  - Local Institution - 2109, Boston, Massachusetts
  - Local Institution - 2106, Ann Arbor, Michigan
  - Local Institution - 2113, Detroit, Michigan
  - Local Institution - 2103, St Louis, Missouri
  - Local Institution - 2104, Toledo, Ohio
  - Local Institution - 2101, Houston, Texas
  - Local Institution - 2112, Fairfax, Virginia
- France (4):
  - Local Institution - 4202, La Tronche, Auvergne-Rhône-Alpes
  - Local Institution - 4203, Saint-Mandé, Val-de-Marne
  - Local Institution - 4204, Villejuif, Val-de-Marne
  - Local Institution - 4201, Lyon
- Local Institution - 6304, Seoul, North Korea
- South Korea (3):
  - Local Institution - 6301, Seoul, Seoul-teukbyeolsi [Seoul]
  - Local Institution - 6303, Seoul
  - Local Institution - 6302, Seoul
- Spain (4):
  - Local Institution - 4104, Madrid
  - Local Institution - 4103, Madrid
  - Local Institution - 4101, Madrid
  - Local Institution - 4102, Pamplona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com